CLINICAL TRIAL: NCT07346742
Title: Intravenous Prophylactic Antibiotics and Antimicrobial-Coated Sutures in Preventing Surgical Site Infection in Open Paediatric Groin Surgeries: A 3-arm Randomized Controlled Trial
Brief Title: Prevention of Surgical Site Infection in Open Paediatric Groin Surgeries Using Intravenous Prophylactic Antibiotics and Antimicrobial-coated Sutures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olawumi Olajide (Other)
Responsible Party: Sponsor-Investigator, Olawumi Olajide, Senior Registrar, Obafemi Awolowo University Teaching Hospital
Organization: Obafemi Awolowo University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ERC/2024/08/11
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inguinal Hernia; Hydroceles; Surgical Site Infection
Keywords: Paediatric groin surgeries; Intravenous prophylactic antibiotics; Antimicrobial-coated sutures; Double blinded randomized controlled trial
MeSH Terms: conditions — Hernia, Inguinal; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- No Antibiotics arm (Placebo Comparator): Participants will have intravenous placebo injection given at the induction of anaesthesia and their surgical wounds closed using non-coated sutures
  Interventions: Other: Placebo intravenous injection
- Intravenous prophylactic antibiotic arm (Active Comparator): Participants will have an intravenous prophylactic antibiotics given at the induction of anaesthesia and their wounds closed with non-coated sutures
  Interventions: Drug: Intravenous Cefuroxime
- Antimicrobial-coated suture arm (Experimental): Participants will have an intravenous placebo injection given at the induction of anaesthesia and their wounds closed with antimicrobial-coated sutures
  Interventions: Device: Antimicrobial-coated sutures

INTERVENTIONS:
Device: Antimicrobial-coated sutures — Use of Antimicrobial-coated sutures to close all layers of the surgical wound following open paediatric groin surgery
  Arms: Antimicrobial-coated suture arm
Drug: Intravenous Cefuroxime — Intravenous cefuroxime is given at the induction of anaesthesia
  Arms: Intravenous prophylactic antibiotic arm
Other: Placebo intravenous injection — 0.2ml of Vitamin Bco injection + 9.8ml sterile water
  Arms: No Antibiotics arm

SUMMARY:
The goal of this clinical trial is to learn if the use of prophylactic antibiotics and antimicrobial-coated sutures can prevent surgical site infection in children undergoing open groin surgeries. The main question it aims to answer is:

• Does the use of intravenous prophylactic antibiotics or antimicrobial-coated sutures significantly reduce the occurrence of surgical site infection in children undergoing open groin surgeries?

Researchers will compare no antibiotic use to the use of intravenous prophylactic antibiotics, or antimicrobial-coated sutures to see if the use of intravenous prophylactic antibiotics and antimicrobial-coated sutures significantly reduces the occurrence of surgical site infection following open groin surgeries in children.

Participants will:

* Undergo open groin surgery with either the use of intravenous prophylactic antibiotic or antimicrobial-coated sutures or without antibiotic use
* Visit the clinic on postoperative days 5, 13 and 30 for review of the surgical wounds for any sign of infection.

DETAILED DESCRIPTION:
The aim of this clinical trial is to learn if the use of intravenous prophylactic antibiotics and antimicrobial-coated sutures can prevent surgical site infection in children undergoing open groin surgeries. The specific objectives are:

* To determine the rate of surgical site infection in paediatric groin surgeries without antibiotics
* To determine the rate of surgical site infection in paediatric groin surgeries with the use of intravenous prophylactic antibiotics
* To determine the rate of surgical site infection in paediatric groin surgeries with the use of antimicrobial-coated sutures.
* To compare the rates of surgical site infection in paediatric groin surgeries without antibiotics, with the use of intravenous prophylactic antibiotics and use of antimicrobial-coated sutures

Researchers will compare no antibiotic use to the use of intravenous prophylactic antibiotics, or antimicrobial-coated sutures to see if the use of intravenous prophylactic antibiotics and antimicrobial-coated sutures significantly reduces the occurrence of surgical site infection following open groin surgeries in children.

It shall be a double blinded randomized controlled trial

Eligible Participants will:

* On the morning of the surgery be randomly assigned to either group A or B or C
* Participants in group A will have intravenous placebo injection given at the induction of anaesthesia and their surgical wounds closed using non-coated sutures
* Participants in group B will have intravenous prophylactic antibiotic given at the induction of anaesthesia and their surgical wounds closed using non-coated sutures
* Participants in group C will have intravenous placebo injection given at the induction of anaesthesia and their surgical wounds closed using antimicrobial-coated sutures
* Visit the clinic on postoperative days 5, 13 and 30 for review of the surgical wounds for any sign of infection following the CDC guidelines.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical conditions requiring daycase open groin surgery

Exclusion Criteria:

1. Re-operations
2. Immunocompromised patients
3. Malnourished patients
4. Complicated groin pathologies e,g obstructed inguinal hernia
5. History of antibiotic usage in the last seven days

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30 days post operative period

CONTACTS AND LOCATIONS:
Locations (1):
- Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No